CLINICAL TRIAL: NCT03794453
Title: Longitudinal Changes in Intestinal Microbiota and Its Association With Acquisition of Antimicrobial Resistance in a Cohort of Stroke Patients
Brief Title: Intestinal Microbiota and Antimicrobial Resistance
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Grace Lui, Assistant Professor, Chinese University of Hong Kong
Other Study IDs: STM_protocol_v1_20180411
Record Dates: First submitted 2019-01-03; First posted 2019-01-07 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Drug Resistance, Microbial
Keywords: Stroke; Intestinal microbiota; Antimicrobial resistance
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool samples for microbiota analysis
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stroke patients

SUMMARY:
Antimicrobial resistance is regarded as one of the major global public health threats, causing at least 700,000 deaths per year. It has been estimated that if the current problem of antimicrobial resistance is not effectively tackled, it would cause the death of 10 million people worldwide by 2050. Multi-drug resistant pathogen is the single most important contributing factor for inappropriate antibiotics therapy, and this in turn lead to higher mortality in patients with sepsis. The slow pace of development of new classes of antimicrobial agents limits the availability of effective therapy for multi-drug resistant organisms, both currently and in the near future. It is therefore of utmost importance to look for strategies to reduce the spread and burden of antimicrobial resistance.

Intestinal microbiota probably played a dominant role in determining the risk of acquisition of multi-drug resistant organisms. For instance, findings from a mouse model showed that Barnesiella species conferred resistance to intestinal colonization by vancomycinresistant Enterococcus. Such findings were subsequently confirmed in human subjects.

This is a prospective longitudinal observational study evaluating the correlation between changes in intestinal microbiota and acquisition of antimicrobial resistance in patients hospitalized for stroke.

Adult patients admitted to the Medical unit of the Prince of Wales Hospital with a diagnosis of acute stroke will be screened for eligibility and will be invited to participate in this study. Data collected from this study will determine the correlation between antibiotics use and changes in intestinal microbiota in a cohort of hospitalized patients as well as the correlation between intestinal microbiota and acquisition of intestinal colonization or infection caused by resistant pathogens.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or above, and
* Radiological evidence of acute ischaemic or hemorrhagic stroke
* Within two days of hospital admission

Exclusion Criteria:

* Use of antibiotics within 4 weeks prior to the time of screening
* Underlying gastrointestinal diseases, including gastrointestinal malignancy, inflammatory bowel disease, resection of small or large bowel
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a diagnosis of acute stroke
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-08-06 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients acquiring intestinal colonization of resistant organisms | 2 years
  Intestinal colonization of resistant organisms are defined as the presence of ESBL or resistance to one or more carbapenems in Enterobacteriaceae identified in the stool samples, in patients without these organisms detected in their stool samples at the time of admission to hospital.

SECONDARY OUTCOMES:
Proportion of patients acquiring nosocomial infections secondary to multi-drug resistant pathogens. | 2 years
  Nosocomial infections are defined as infections with onset of 72 hours or more after hospital admission.
  Multi-drug resistant pathogens are defined as methicillin-resistant Staphylococcus aureus, vancomycin-resistant Enterococcus species, ESBL-producing Enterobacteriaceae, and carbapenem-resistant Gram-negative bacteria, including Enterobacteriaceae, Acinetobacter species, and Pseudomonas aeruginosa, detected in one or more of patients' clinical specimens.

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided